CLINICAL TRIAL: NCT00363558
Title: Fixation of Skin Grafts in Patients With Burns: Comparison Between Cyanoacrylate Glue and Skin Staples
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Other Study IDs: 4133
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2003-05

CONDITIONS: Grafting, Skin; Burn
Keywords: skin graft; fixation; cyanoacrylate glue; skin staples
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Retrospective

SUMMARY:
Skin graft fixation is essential for the success of its survival. There are several common methods for skin graft fixation including sutures, skin staples and glue. The study objective is to compare between skin graft fixation with staples and glue in burn patients. The study is retrospective. It Includes 44 patients that were hospitalized in the burn unit, Rabin Medical Center, Israel with 2nd and 3rd degree burns, total body surface area 1-50% during 1/2002-5/2003.All patients were operated for debridement and skin grafting. In 29 patients the skin graft was fixated with staples and in 15 with cyanoacrylate glue (histoacryl). The parameters that will be compared are skin graft take, hospitalization length and local infection.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with 2nd and 3rd degree burns who were operated for debridement and skin grafting
* burn total body surface area 1-50%

Exclusion Criteria:

* burn total body surface area> 50%

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44
Dates: Start 2002-01; Study Completion 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Neta Adler, MD, Principal Investigator — Rabin Medical Center , Israel
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Kaplan HY. A quick stapler tie-over fixation for skin grafts. Ann Plast Surg. 1989 Feb;22(2):173-4. doi: 10.1097/00000637-198902000-00015. PMID 2660713
- [Background] Zaki I, Scerri L, Millard L. Split skin grafting on severely damaged skin. A technique using absorbable tissue adhesive. J Dermatol Surg Oncol. 1994 Dec;20(12):827-9. doi: 10.1111/j.1524-4725.1994.tb03713.x. PMID 7798416
- [Background] Shorr N, Cohen MS, Lessner A. Histoacryl closure of eyelid skin grafts. Ophthalmic Plast Reconstr Surg. 1991;7(3):190-3. doi: 10.1097/00002341-199109000-00007. PMID 1911525